CLINICAL TRIAL: NCT00533702
Title: Phase II Randomized, Open-Label Study of IMC-1121B With or Without Dacarbazine in Patients With Metastatic Malignant Melanoma
Brief Title: A Study of IMC-1121B (Ramucirumab) With or Without Dacarbazine in Metastatic Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13920; CP12-0604 (Other: ImClone Systems); I4T-IE-JVBO (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-09-17; First posted 2007-09-21 (Estimated); Results first posted 2014-06-18 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Metastatic Malignant Melanoma
Keywords: Phase II; Melanoma; IMC-1121B; ImClone
MeSH Terms: conditions — Melanoma | interventions — Ramucirumab; Dacarbazine; imidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMC-1121B (ramucirumab) (Experimental): IMC-1121B (ramucirumab)
  Interventions: Biological: IMC-1121B (ramucirumab)
- IMC-1121B (ramucirumab) + dacarbazine (Active Comparator): IMC-1121B (ramucirumab) + dacarbazine
  Interventions: Biological: IMC-1121B (ramucirumab); Drug: Dacarbazine

INTERVENTIONS:
Biological: IMC-1121B (ramucirumab) — 10 milligrams/kilogram (mg/kg) intravenously every 3 weeks in the absence of disease progression, unacceptable toxicity, or other withdrawal criteria.
  Other Names: ramucirumab; LY3009806
Drug: Dacarbazine — 1000 milligrams/square meter (mg/m2) intravenously every 3 weeks in the absence of disease progression, unacceptable toxicity, or other withdrawal criteria.
  Other Names: DIC; Imidazole; Carboxamide
  Arms: IMC-1121B (ramucirumab) + dacarbazine

SUMMARY:
The primary objective of this study is to determine the progression-free survival (PFS) of participants with previously untreated metastatic malignant melanoma when treated with IMC-1121B (ramucirumab) alone or in combination with dacarbazine.

DETAILED DESCRIPTION:
The purpose of this study is to determine the antitumor activity and safety profile of IMC-1121B (ramucirumab) when used alone or in combination with dacarbazine in participants with metastatic melanoma who have not received prior chemotherapy for this disease.

ELIGIBILITY:
Inclusion Criteria:

* The participant has histologically or cytologically confirmed melanoma that is stage IV (metastatic)
* The participant has an Eastern Cooperative Oncology Performance Status (ECOG PS) of 0-1
* The participant has completed any prior radiotherapy, biologic/immunotherapy or vaccine therapy (for adjuvant or advanced disease) at least six weeks prior to the first dose of study therapy
* The participant has adequate hematological functions [absolute neutrophil count (ANC) ≥ 1500 cells/microliter (μL), hemoglobin ≥ 9 grams/deciliter (g/dL) and platelets ≥ 100,000 cells/μL].
* The participant has adequate hepatic function [bilirubin within normal limits (WNL), aspartate transaminase (AST) and/or alanine transaminase (ALT) ≤ 2.5 times the upper limit of normal (ULN), or ≤ 5.0 times the ULN if the transaminase elevation is due to liver metastases]
* The participant has serum creatinine ≤ 1.5 x ULN [or a calculated creatinine clearance > 60 milliliters/minute (mL/min)]
* The participant's urinary protein ≤ 1+ on dipstick or routine urinalysis [(UA); if urine dipstick or routine analysis is ≥ 2+, a 24-hour urine for protein must demonstrate < 1000 milligrams (mg) of protein in 24 hours to allow participation in the study]
* The participant must have adequate coagulation function as defined by International Normalized Ratio (INR) ≤ 1.5 and a partial thromboplastin time (PTT) ≤ 1.5 X ULN

Exclusion Criteria

* The participant has mucosal or intra-ocular melanoma
* The participant has known or suspected brain or leptomeningeal metastases
* The participant has had prior cytotoxic chemotherapy for metastatic malignant melanoma
* The participant has had more than one line of biologic, immunologic or vaccine-based therapy for metastatic malignant melanoma (including therapy for adjuvant or advanced disease)
* The participant has a nonhealing wound or ulcer
* The participant has a known alcohol or drug dependency
* The participant is pregnant or breastfeeding
* The participant has a coexisting medical or psychiatric problem of sufficient severity to limit compliance with the study and/or increase the risks associated with study participation or study drug administration or interfere with the interpretation of study results
* The participant has an ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, psychiatric illness/social situations, or any other serious uncontrolled medical disorders in the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2007-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (15):
- United States (15):
  - ImClone Investigational Site, Decatur, Alabama
  - ImClone Investigational Site, Scottsdale, Arizona
  - ImClone Investigational Site, Fresno, California
  - ImClone Investigational Site, San Francisco, California
  - ImClone Investigational Site, Aurora, Colorado
  - ImClone Investigational Site, Jacksonville, Florida
  - ImClone Investigational Site, Orlando, Florida
  - ImClone Investigational Site, Oxford, Mississippi
  - ImClone Investigational Site, Missoula, Montana
  - ImClone Investigational Site, Buffalo, New York
  - ImClone Investigational Site, New York, New York
  - ImClone Investigational Site, Willow Grove, Pennsylvania
  - ImClone Investigational Site, Dallas, Texas
  - ImClone Investigational Site, Houston, Texas
  - ImClone Investigational Site, Seattle, Washington

REFERENCES:
- [Derived] Carvajal RD, Wong MK, Thompson JA, Gordon MS, Lewis KD, Pavlick AC, Wolchok JD, Rojas PB, Schwartz JD, Bedikian AY. A phase 2 randomised study of ramucirumab (IMC-1121B) with or without dacarbazine in patients with metastatic melanoma. Eur J Cancer. 2014 Aug;50(12):2099-107. doi: 10.1016/j.ejca.2014.03.289. Epub 2014 Jun 12. PMID 24930625

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed the study were those who died or were alive but off treatment at the end of the study.
Groups:
- IMC-1121B (Ramucirumab) + Dacarbazine: IMC-1121B (ramucirumab): 10 milligrams/kilogram (mg/kg) administered intravenously on Day 1 of 21-day cycle in the absence of disease progression, unacceptable toxicity, or other withdrawal criteria.
  Dacarbazine: 1000 milligrams/square meter (mg/m2) administered intravenously on Day 1 of 21-day cycle in the absence of disease progression, unacceptable toxicity, or other withdrawal criteria.
- IMC-1121B (Ramucirumab): IMC-1121B (ramucirumab): 10 mg/kg administered intravenously on Day 1 of 21-day cycle in the absence of disease progression, unacceptable toxicity, or other withdrawal criteria.
Period: Overall Study
Arm/Group | IMC-1121B (Ramucirumab) + Dacarbazine | IMC-1121B (Ramucirumab)
Started | 54 | 52
Received Any Quantity of Study Drug | 52 | 50
Completed | 49 | 50
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Found ineligible after randomization | 2 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who were treated with any quantity of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | IMC-1121B (Ramucirumab) + Dacarbazine | IMC-1121B (Ramucirumab) | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 28 | 57
  >=65 years | 23 | 22 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 12 | 27
  Male | 37 | 38 | 75
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 47 | 49 | 96
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 52 | 50 | 102
Race [Number; unit: participants]
  Asian | 1 | 0 | 1
  White | 50 | 50 | 100
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the time from the first day of therapy to the first evidence of disease progression as defined by Response Evaluation Criteria in Solid Tumors (RECIST v1.0) or death from any cause. Progressive disease (PD) was defined as at least a 20% increase in the sum of the longest diameter (LD) of the target lesions, taking as reference the smallest sum LD recorded since the treatment started in comparison with the measurement of the nadir or the appearance of 1 or more new lesions. In addition, unequivocal progression of existing non-target lesions was considered PD. New or existing pleural effusion/ascites required cytological confirmation for PD according to the protocol. Participants who did not progress and who were alive or did not have documented progression or missed ≥2 visits, or had no post baseline assessment were censored at the day of their last tumor assessment.
Time Frame: Baseline up to 36 months
Population: Intent-to-Treat Population: All enrolled participants who were treated with any quantity of study drug. Censored participants: IMC-1121B (ramucirumab) + dacarbazine=9; IMC-1121B (ramucirumab)=4.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-1121B (Ramucirumab) + Dacarbazine | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 52 | 50
months | 2.6 [1.4 to 5.4] | 1.7 [1.4 to 2.9]

2. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: The number of participants who experienced any IMC-1121B (ramucirumab [RAM]) treatment-related and treatment emergent AE (TEAE), treatment-related TEAE of Grade ≥3, treatment-related TE serious AEs (SAEs), treatment-related TEAE resulting in death (Grade 5 AE) and any TEAEs resulting in death. A summary of SAEs and all other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to 40 months
Population: Safety Population: All enrolled participants who were treated with any quantity of study drug.
Measure: Number; unit: participants
Arm/Group | IMC-1121B (Ramucirumab) + Dacarbazine | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 52 | 50
participants
  Any RAM related TEAE | 43 | 40
  RAM related SAE | 9 | 5
  RAM related ≥ Grade 3 AE | 20 | 13
  RAM related death | 1 | 1
  RAM related TEAE leading to discontinuation of RAM | 3 | 4
  Any AE with outcome of death | 2 | 2

3. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) [Overall Response Rate (ORR)]
Description: The ORR was defined as the percentage of all randomized participants with the best overall response of PR or CR using Response Evaluation Criteria in Solid Tumors (RECIST v1.0). CR was defined as the disappearance of all target and non-target lesions. PR was defined as at least a 30% decrease in sum of longest diameter of target lesions. CR and PR had to be confirmed by repeat assessments and performed no fewer than 4 weeks after the criteria for response were first met.
Time Frame: Cycle 1 Day 1 (of 21-day cycle) up to 17.1 months
Population: Intent-to-Treat Population: All enrolled participants who were treated with any quantity of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | IMC-1121B (Ramucirumab) + Dacarbazine | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 52 | 50
percentage of participants | 17.3 [8.2 to 30.3] | 4.0 [0.5 to 13.7]

4. Secondary Outcome: Duration of Response
Description: The duration of overall response was defined as the time from first assessment of complete response (CR) or partial response (PR) to the first date of progressive disease (PD) using Response Evaluation Criteria in Solid Tumors (RECIST v1.0), initiation of other or additional antitumor therapy, or death from any cause. CR was defined as the disappearance of all target lesions. PR was defined as having at least a 30% decrease in sum of longest diameter of target lesions. CR and PR had to be confirmed by repeat assessments and performed no fewer than 4 weeks after the criteria for response were first met. PD was defined as at least 20% increase in sum of longest diameter of target lesions. Participants who did not relapse were censored at the day of their last objective tumor assessment.
Time Frame: Cycle 1 Day 1 (of 21-day cycle) up to 17.1 months
Population: Intent-to-Treat Population: All enrolled participants who were treated with any quantity of study drug and who had CR or PR. Censored participants: IMC-1121B (ramucirumab) + dacarbazine=2; IMC-1121B (ramucirumab)=0.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | IMC-1121B (Ramucirumab) + Dacarbazine | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 9 | 2
months | 11.0 [3.9 to 17.1] | NA [3.2 to 14.0] — Median was not calculated since there are only 2 data points.

5. Secondary Outcome: Percentage of Participants With Stable Disease (SD) or Better (Disease Control Rate) at 6 Weeks
Description: Disease Control Rate (DCR) was defined as complete response (CR) plus partial response (PR) plus SD using Response Evaluation Criteria in Solid Tumors (RECIST v1.0). CR was defined as the disappearance of all target and non-target lesions and the normalization of non-target lesion tumor marker levels. PR was defined as at least a 30% decrease from baseline in sum of longest diameter of target lesions. CR and PR had to be confirmed by repeat assessments and performed no fewer than 4 weeks after the criteria for response were first met. SD was defined as: neither sufficient increase to qualify for progressive disease (PD) nor sufficient shrinkage to qualify for PR, taking as reference the smallest sum of the longest diameters recorded since treatment began. PD was defined as at least 20% increase in sum of longest diameter of target lesions.
Time Frame: 6 weeks (2 cycles of treatment)
Population: Intent-to-Treat Population: All enrolled participants who were treated with any quantity of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | IMC-1121B (Ramucirumab) + Dacarbazine | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 52 | 50
percentage of participants | 54 | 44

6. Secondary Outcome: Percentage of Participants With Stable Disease (SD) or Better (Disease Control Rate) at 12 Weeks
Description: Disease Control Rate (DCR) was defined as complete response (CR) plus partial response (PR) plus SD using Response Evaluation Criteria in Solid Tumors (RECIST v1.0). CR was defined as the disappearance of all target and non-target lesions and the normalization of non-target lesion tumor marker levels. PR was defined as at least a 30% decrease from baseline in sum of longest diameter of target lesions. CR and PR had to be confirmed by repeat assessments and performed no fewer than 4 weeks after the criteria for response were first met. Stable Disease (SD) was defined as: neither sufficient increase to qualify for progressive disease (PD) nor sufficient shrinkage to qualify for PR, taking as reference the smallest sum of the longest diameters recorded since treatment began. PD was defined as at least 20% increase in sum of longest diameter of target lesions.
Time Frame: 12 weeks (4 cycles of treatment)
Population: Intent-to-Treat Population: All enrolled participants who were treated with any quantity of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | IMC-1121B (Ramucirumab) + Dacarbazine | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 52 | 50
percentage of participants | 40 | 24

7. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Response Rate) at 12 Weeks
Description: Response rate was defined as a CR or a PR using Response Evaluation Criteria in Solid Tumors (RECIST v1.0). CR was defined as the disappearance of all target and non-target lesions and the normalization of non-target lesion tumor marker levels. PR was defined as at least a 30% decrease from baseline in sum of longest diameter of target lesions. CR and PR had to be confirmed by repeat assessments and performed no fewer than 4 weeks after the criteria for response were first met.
Time Frame: 12 weeks (4 cycles of treatment)
Population: Intent-to-Treat Population: All enrolled participants who were treated with any quantity of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | IMC-1121B (Ramucirumab) + Dacarbazine | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 52 | 50
percentage of participants | 13.5 | 4.0

8. Secondary Outcome: Maximum Concentration (Cmax) for Cycle 1 Day 1
Description: Cmax was not calculated due to sparse sampling.
Time Frame: Cycle 1 Day 1 (21-day cycle) 1-hour post infusion
Population: Zero participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab) + Dacarbazine | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Maximum Concentration (Cmax) for Cycle 1 Day 7
Description: Cmax was not calculated due to sparse sampling.
Time Frame: Cycle 1 Day 7 (21-day cycle)
Population: Zero participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab) + Dacarbazine | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Maximum Concentration (Cmax) for Cycle 1 Day 14
Description: Cmax was not calculated due to sparse sampling.
Time Frame: Cycle 1 Day 14 (21-day cycle)
Population: Zero participants were analyzed.
Arm/Group | IMC-1121B (Ramucirumab) + Dacarbazine | IMC-1121B (Ramucirumab)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | IMC-1121B (Ramucirumab) + Dacarbazine | IMC-1121B (Ramucirumab)
Serious Adverse Events (participants affected / at risk) | 14/52 | 15/50
Other Adverse Events (participants affected / at risk) | 52/52 | 48/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-1121B (Ramucirumab) + Dacarbazine (N=52) | IMC-1121B (Ramucirumab) (N=50)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) — Event resulted in death
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 3 (3)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 2 (3) — Event resulted in death in both participants
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Event resulted in death
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IMC-1121B (Ramucirumab) + Dacarbazine (N=52) | IMC-1121B (Ramucirumab) (N=50)
Anaemia (Blood and lymphatic system disorders) | 7 (22) | 2 (4)
Leukopenia (Blood and lymphatic system disorders) | 5 (15) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 18 (29) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 20 (54) | 4 (7)
Vision blurred (Eye disorders) | 1 (1) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 16 (23) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 10 (13) | 8 (10)
Dry mouth (Gastrointestinal disorders) | 4 (5) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gingival bleeding (Gastrointestinal disorders) | 3 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 20 (36) | 14 (19)
Vomiting (Gastrointestinal disorders) | 7 (9) | 11 (12)
Chest pain (General disorders) | 3 (3) | 2 (2)
Chills (General disorders) | 6 (7) | 8 (8)
Fatigue (General disorders) | 33 (63) | 28 (38)
Infusion related reaction (General disorders) | 4 (4) | 4 (5)
Infusion site pain (General disorders) | 3 (3) | 0 (0)
Injection site irritation (General disorders) | 4 (8) | 0 (0)
Oedema peripheral (General disorders) | 15 (27) | 10 (12)
Pain (General disorders) | 4 (4) | 2 (2)
Pyrexia (General disorders) | 2 (3) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 6 (7) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 5 (12)
Anorexia (Metabolism and nutrition disorders) | 14 (15) | 7 (8)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (10) | 9 (14)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (7) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2)
Dizziness (Nervous system disorders) | 3 (5) | 2 (2)
Dysgeusia (Nervous system disorders) | 5 (6) | 3 (3)
Headache (Nervous system disorders) | 9 (18) | 16 (21)
Paraesthesia (Nervous system disorders) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 5 (6) | 4 (4)
Depression (Psychiatric disorders) | 4 (4) | 4 (4)
Insomnia (Psychiatric disorders) | 9 (9) | 5 (5)
Dysuria (Renal and urinary disorders) | 0 (0) | 4 (5)
Proteinuria (Renal and urinary disorders) | 4 (8) | 6 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 5 (7)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 4 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 (12) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (10) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 8 (12) | 8 (11)
Vitiligo (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Flushing (Vascular disorders) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 12 (18) | 12 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.